CLINICAL TRIAL: NCT04231253
Title: T Cell/B Cell Collaboration in Multiple Sclerosis: Exploring an Intimate Relationship
Brief Title: MUltiple Sclerosis : T Cell / B Cell Exploration
Acronym: MUST-BE
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_8871_MUST-BE
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study, an ancillary to ABCD-SEP (NCT03744351), will be interested in more precisely characterizing circulating and infiltrating TH cells in Multiple Sclerosis whether at the transcriptomic level or at the functional level.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory demyelinating disease of the Central Nervous System (CNS) affecting mostly young adults between 20 and 40 years of age. This disease is the leading cause of non-traumatic disability in young adults.

MS has long been considered a predominantly T-cell mediated disease. However, the remarkable efficacy of anti-CD20 monoclonal antibodies in this disease has demonstrated the major role of B-cell in the pathophysiology of this disease.

The B-cell have many functions: these cells are indeed able to secrete cytokines (pro and anti inflammatory), to present antigens to T lymphocytes, but also to differentiate into plasmocytic cells and thus to secrete immunoglobulins. Several studies have shown that B-cell in patients with MS secrete significantly more pro-inflammatory cytokines (GM-CSF, IL-6, TNFα). In addition, infiltrates and tertiary lymphoid structures have been found in the meninges of patients with MS, particularly in progressive forms of the disease. It seems clear to this day that these cells are strongly involved in the development of MS. Despite the many advances made recently in understanding the role of B-cell in the pathophysiology of MS, the precise involvement of plasma cells and their functions at different stages of the disease remains unclear.

Folluclar helper T cells (TFH) play a crucial role in lymphocyte B differentiation. These cells are located within the germinal centers in the secondary lymphoid organs, and their memory compartment also circulates in the blood. Several circulating TFH subpopulations have recently been defined, with different "helping" capacities.

This study, an ancillary to ABCD-SEP (NCT03744351), will be interested in more precisely characterizing circulating and infiltrating TH cells in Multiple Sclerosis whether at the transcriptomic level or at the functional level.

ELIGIBILITY:
Inclusion Criteria:

Regarding MS patients (remitting or progressive untreated):

* Adult (age greater than or equal to 18 years) of both sexes;
* MS fulfilling the criteria of McDonald 2017;
* Remittent or progressive form;
* No immunomodulatory or immunosuppressive therapy for at least 3 months;
* Free, informed and written consent signed by the patient.

Regarding Clinically Isolated Syndrome:

* Adult (age greater than or equal to 18 years) of both sexes;
* Clinically isolated syndrome suggestive of MS (at least two typical lesions in two different locations);
* Patient receiving a Lumbar Puncture (PL) for diagnostic purposes;
* No immunomodulatory or immunosuppressive therapy for at least 3 months;
* Free, informed and written consent signed by the patient.

Regarding non-MS patients with neurological inflammatory disease:

* Adult (age greater than or equal to 18 years) of both sexes;
* Patient with non-MS neurological inflammatory disease (examples: meningitis, neurolupus, neurosarcoidosis...);
* Patients with PL for diagnostic or surveillance purposes;
* No immunomodulatory or immunosuppressive therapy for at least 3 months;
* Free, informed and written consent signed by the patient.

Regarding healthy volunteers:

* Adult (age greater than or equal to 18 years) of both sexes;
* Free, informed and written consent signed by the volunteer.

Exclusion Criteria:

Regarding all patients:

* Pregnancy;
* Breastfeeding;
* Treatment with corticotherapy in the last month;
* Patient not affiliated to health insurance;
* Persons major subject to legal protection (safeguard of justice, guardianship, tutorship), persons deprived of their liberty.

Regarding healthy volunteers:

* Pregnancy;
* Breastfeeding;
* Not affiliated to social security;
* Persons major subject to legal protection (safeguard of justice, guardianship, tutorship), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population concerned is the same as the one participating in the ABCD-SEP study.
  These patients gave their consent for the remaining biological samples to be used for ulterior research
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
To compare the transcriptome profile of infiltrating TFH cells from CIS patients to non-MS patients with neurological inflammatory diseases | At inclusion
  Comparison of each gene expression of infiltrating TFH cells from CIS patients to those of non-MS patients with neurological inflammatory diseases by RNAsequencing

SECONDARY OUTCOMES:
To compare the transcriptome profile of infiltrating TFH cells from CIS patients to healthy volunteers. | At inclusion
  Comparison of each gene expression of infiltrating TFH cells from CIS patients to those of healthy volunteers (HV) by RNAsequencing
To compare the B cell differentiation helping abilities of TFH cells from MS patients to those of HV | At inclusion
  Analysis of B cell phenotype after 7 days of in vitro coculture assays and comparison of the frequencies between MS patients and HV
To compare the migration abilities of TFH cells from MS patients to those of HV | At inclusion
  Analysis of the rate, number and phenotype of migrating TFH cells after 12 to 24 hours using an in vitro model of Blood Brain Barrier in MS patients compared to HV

CONTACTS AND LOCATIONS:
Overall Officials: Laure Michel, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France